CLINICAL TRIAL: NCT05991115
Title: The Hospital to Home Study: a Pragmatic Trial to Optimize Transitions and Address Disparities in Asthma Care
Brief Title: Hospital to Home Study: Trial to Optimize Transitions and Address Disparities in Asthma Care
Acronym: H2H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kavita Parikh (Other)
Responsible Party: Sponsor-Investigator, Kavita Parikh, Associate Professor of Pediatrics, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY0699
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Asthma; Asthma in Children
Keywords: asthma; hospitalization; children
MeSH Terms: conditions — Asthma | interventions — Hospital to Home Transition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Control arm will receive the standard of care (SOC) after hospital discharge.
- Hospital to Home Transition (H2H) (Experimental): The intervention for this study is a multi-component navigation-supported intervention for children hospitalized with asthma. Navigators will work with families for 12-months post-discharge. Trained asthma educator/navigators will work to address challenges with asthma care after discharge; will include maximum 15 contacts/12 months. The asthma navigators within this study will attempt to maintain direct contact with participants primary care doctors through email, fax, and/or postal mail as means for delivering asthma action plans, prescription updates, and patient appointment scheduling. The asthma navigators for intervention participants will attempt to maintain contact with the school nurse in efforts to have a line of communication with the school. Asthma navigators will assist families in all home-based needs pertaining to their child's asthma.
  Interventions: Behavioral: Hospital to Home Transition (H2H)

INTERVENTIONS:
Behavioral: Hospital to Home Transition (H2H) — The intervention for this study is a multi-component navigation-supported intervention for children hospitalized with asthma. Navigators will work with families for 12-months post-discharge. Trained asthma educator/navigators will work to address challenges with asthma care after discharge; will include maximum 15 contacts/12 months. The asthma navigators within this study will attempt to maintain direct contact with participants primary care doctors through email, fax, and/or postal mail as means for delivering asthma action plans, prescription updates, and patient appointment scheduling. The asthma navigators for intervention participants will attempt to maintain contact with the school nurse in efforts to have a line of communication with the school. Asthma navigators will assist families in all home-based needs pertaining to their child's asthma.
  Arms: Hospital to Home Transition (H2H)

SUMMARY:
Caregiver-child dyads will be recruited during child's hospital admission for asthma exacerbation. Recruitment sites will be mainly Children's National Hospital Sheikh Zayed campus, as well as regional partners: Holy Cross Hospital, and Mary Washington Hospital. After enrollment, baseline data will be collected from caregiver. Caregiver-child dyads will be randomized (1:1 ratio) into the control arm or intervention arm. Control arm will receive the standard of care after hospital discharge. Intervention arm will receive the SOC plus an asthma navigator support after hospital discharge. Caregivers in both arms will complete data collection surveys (either in-person or via telehealth) at 3-,6-, 9-, and 12- month post enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. speak English or Spanish
2. are at least 18 years old
3. live in the District of Columbia, Maryland, or Virginia (DMV)
4. have a child aged 4-12 years who is hospitalized due to asthma exacerbation.

Exclusion Criteria:

1. . Children ages 4-12 years with chronic medical condition (other than asthma) including but not limited to diabetes, sickle cell disease, heart disease, lung disease or neurological disorder
2. . Children ages 4-12 years involved in interventions with behavioral component and/or novel asthma therapeutics will be excluded given overlap with the current intervention
3. . Children ages 4-12 years in foster care
4. . Families not residing in the DMV
5. . Caregivers who do not speak English or Spanish

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 340 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Re-admissions | 3, 6, 9, 12 months
  Asthma-related readmissions over 12-month follow-up period from index hospitalization

SECONDARY OUTCOMES:
Number of Emergency Department (ED) Visit | 3, 6, 9, 12 months
  Asthma-related ED visits over 12-month follow-up period from index hospitalization
Asthma Control Test (ACT) | 3, 6, 9, 12 months
  Asthma Control Test (ACT) which is 7 questions with scores ranging from 0 to 27. Score less than 19 means that asthma is not well-controlled.
Number of Household Triggers | 3, 6, 9, 12 months
  Questionnaire from home visit program. Includes exposures in the home, specifically: birds, cats, dogs, dust, eats in Bedroom, tobacco smoke, fireplace/wood burning stove/heat source, incense/candles, mice/rats, roaches/waterbugs, mold/mildew smell;water damage, perfume, other.
Caregiver quality of life | 3 ,6, 9, 12 months
  Pediatric Asthma Caregivers Quality of Life Questionnaire (PACQLQ) which includes 13-items; includes feelings about child's asthma symptoms (9 items), level of concern about child's asthma (4 items); uses a 7-point Likert scale.Responses to each item of the PACQLQ are given on a seven-point scale, ranging from 1 to 7, with the higher scores indicating less impairment. The result will be expressed as a mean score per item for each of the domains, as well as for the overall quality of life. Higher score means better outcome.
Symptom Free Days (SFD) | 3, 6, 9, 12 months
  Symptom Free Days (SFD) is measured over the last 14 days, and ranges from 0 to 14. SFD question will be asked at 3,6,9,12 month data collection with a 14 day look-back period.
Parent Self-Efficacy | 3, 6, 9, 12 months
  Parent Asthma Management Self- Efficacy Scale (PAMES) survey includes 13-item questions that measures parent self-efficacy with child's asthma; uses a 5-point scale. Scores range from 13-65. Parents rated their responses on a 5-point ordinal scale from 1= not at all sure to 5 = completely sure. Higher score means better outcome.
Caregiver Stress | 3, 6, 9, 12 months
  Perceived Stress Scale (PSS) is a validated tool with a shorter validated version that can be used for data collection over the phone and uses a 5-point ordinal scale. Individual scores on the PSS can range from 0 to 40 with higher score indicating higher perceived stress. Higher score means worse outcome.
Parental Resilience | 3, 6, 9, 12 months
  Brief Resilience Scale (BRS) is 6-item tool to measure resilience or the ability to bounce back or recover from stress that would be valuable in coping with health-related stressors. Total score will range from 6-30. Higher score means better outcome.

OTHER OUTCOMES:
Sociodemographic factors | Baseline
  Age, Gender, Martial Status, Race, Ethnicity, Socioeconomic status, Occupation, Education, Household size, Number of asthma caregivers, English Proficiency, and Health Literacy
Experience with Discrimination (EOD) | Baseline
  Survey includes experiences with discrimination and situations of unfair treatment asking about frequency as well as the specific situation. Validated close-format questions used in diverse racial/ethnic groups.
Asthma severity | Baseline
  Asthma severity will be measured by NIH classification of Intermittent, Persistent mild, Persistent moderate, Persistent severe.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Parikh, MD MSHS, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States